CLINICAL TRIAL: NCT05072262
Title: A Randomized Clinical Two-arm Trial Comparing Inflammation and Cystoid Macular Edema for the Medication Regimens Postoperative Topical NSAIDs and Steroids to Only Postoperative Topical Steroids in Patients Undergoing Corneal Endothelial Transplantations (DMEC)
Brief Title: DSAEK/DMEK and Cystoid Macular Edema - the Role for Topical NSAIDs (Nepafenac) (DMEC)
Acronym: DMEC
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Olav Kristianslund, Principal investigator, Senior consultant MD PhD, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 131128; 2020-003408-15 (EudraCT Number)
Record Dates: First submitted 2021-09-24; First posted 2021-10-08 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Descemet Stripping Automated Endothelial Keratoplasty (DSAEK); Descemet Membrane Endothelial Keratoplasty (DMEK)

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (dexamethasone only) (Active Comparator): Topical dexamethasone 1 mg/ml (Spersadex) started the day after surgery
  Interventions: Drug: Dexamethasone Ophthalmic
- Study group (NSAIDs and dexamethasone) (Experimental): Topical nepafenac (Nevanac) 3 mg/ml and dexamethasone 1 mg/ml (Spersadex) started the day after surgery.
  Interventions: Drug: Nepafenac Ophthalmic; Drug: Dexamethasone Ophthalmic

INTERVENTIONS:
Drug: Nepafenac Ophthalmic — Topical nepafenac (Nevanac) 3 mg/ml
  Arms: Study group (NSAIDs and dexamethasone)
Drug: Dexamethasone Ophthalmic — Topical dexamethasone 1 mg/ml (Spersadex)

SUMMARY:
The DMEC trial is a randomized clinical two-arm trial comparing inflammation and cystoid macular edema for the medication regimens postoperative topical NSAIDs and steroids to only postoperative topical steroids in patients undergoing corneal endothelial transplantations (DSAEK or DMEK).

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18 years and older at the time of the signing of the informed consent. There is no upper age limit.
* Scheduled for DSAEK or DMEK
* Ability to cooperate fairly well during the examinations
* Willing to participate in the study and capable of giving informed consent, which includes compliance with the requirements and restrictions in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

* Contraindications for use of any medication (as listed in the approved SPC, e.g. allergy, pregnancy, breastfeeding)
* Pregnancy or possible pregnancy during the study period
* Preoperative macular edema and/or ongoing treatment for macular edema
* Re-transplantation
* In-operated glaucoma shunt / valve (e.g. Ahmed glaucoma valve)
* Aphakic eyes (eyes without a biological or artificial intraocular lens)
* Loss of central vision (expected visual acuity potential after surgery below 0.1 Snellen)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-11-25 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Central macular thickness after 4 weeks | 4 weeks after surgery
  Measure central macular thickness (in um) on optical coherence tomography (OCT)
Cystoid macular edema (CME) after 4 weeks | 4 weeks after surgery
  Determine if the patient has CME based on evaluation of macular cysts on optical coherence tomography (OCT)

SECONDARY OUTCOMES:
Intraocular inflammation | Preoperatively, and 1 week, 4 weeks, 2 months and 2 years after surgery
  Measured by laser flare meter
Intraocular pressure | Preoperatively, and 1 day, 1 week, 4 weeks, 2 months and 2 years after surgery
  Measured by tonometry
Visual outcome | Preoperatively, and 1 week, 4 weeks, 2 months and 2 years after surgery
  Measure uncorrected and corrected distance visual acuity using visual acuity chart
Corneal endothelial status | 1 week, 4 weeks, 2 months and 2 years after surgery
  Measure corneal endothelial cell density using microscopy instrument
Patient reported outcome measure (PROM) | 1 week, 4 weeks and 2 months after surgery
  COMToL questionnaire for ocular medication
Central macular thickness (CMT) | Preoperatively, and 1 week, 2 months, and 2 years after surgery
  Measure CMT (in um) on optical coherence tomography (OCT)
Cystoid macular edema (CME) | Preoperatively, and 1 week, 2 months, and 2 years after surgery
  Determine if the patient has CME based on evaluation of macular cysts on optical coherence tomography (OCT)

CONTACTS AND LOCATIONS:
Overall Officials: Olav Kristianslund, MD PhD, Principal Investigator — Department of Ophthalmology, Oslo University Hospital
Locations (1):
- Department of Ophthalmology, Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided